CLINICAL TRIAL: NCT04403802
Title: IIT2019-08-ASHER-VOXXSOCK Voxx Human Performance Technology Socks for Chemotherapy-Induced Peripheral Neuropathy: A Double Blind, Randomized, Controlled Crossover Trial
Brief Title: Voxx Human Performance Technology Socks for Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arash Asher, MD (Other)
Collaborators: VoxxLife (Unknown)
Responsible Party: Sponsor-Investigator, Arash Asher, MD, Director, Cancer Rehabilitation & Survivorship, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IIT2019-08-ASHER-VOXXSOCK
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Neuropathy;Peripheral; Chemotherapy-induced Peripheral Neuropathy; Neuropathy
Keywords: Chemo-induced Peripheral Neuropathy; Voxx Socks; Voxx Human Performance Technology; Voxx HPT
MeSH Terms: conditions — Neuritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Arm A: Voxx socks followed by placebo socks (Experimental): Continuous wear of Voxx Human Performance Technology Socks for 2 weeks, followed by continuous wear of placebo socks for 2 weeks (separated by a 2-week washout period)
  Interventions: Device: Voxx Human Performance Technology Socks; Device: Placebo Socks
- Arm B: Placebo socks followed by Voxx socks (Experimental): Continuous wear of placebo socks for 2 weeks, followed by continuous wear of Voxx Human Performance Technology Socks for 2 weeks (separated by a 2-week washout period)
  Interventions: Device: Voxx Human Performance Technology Socks; Device: Placebo Socks

INTERVENTIONS:
Device: Voxx Human Performance Technology Socks — Voxx Human Performance Technology Socks are commercially-available socks that are drug and electrical free. The Voxx Human Performance Technology proprietary pattern is woven into a sock that is made of 70% cotton, 25% polyester, 3% spandex, and 2% nylon.
  Prior to the 2-week treatment window, patients will be provided with 6 pairs of Voxx Human Performance Technology socks. Patients will be asked to wear the socks continuously during both waking and sleeping hours, except when showering, bathing, or swimming.
Device: Placebo Socks — Placebo socks are identical to the Voxx Human Performance Technology socks but do not include the Voxx Human Performance Technology pattern woven into the sock. Placebo socks are made of the same fabric as Voxx Human Performance Technology socks and are drug and electrical free.
  Prior to the 2-week treatment window, patients will be provided with 6 pairs of placebo socks. Patients will be asked to wear the socks continuously during both waking and sleeping hours, except when showering, bathing, or swimming.

SUMMARY:
This is a double blind, randomized, crossover pilot study of Voxx Human Performance Technology Socks versus placebo socks for the treatment of chemotherapy-induced peripheral neuropathy in patients with cancer. Patients will be randomized 1:1 to one of the following regimens:

* Arm A: Continuous wear of Voxx Human Performance Technology Socks for 2 weeks, followed by continuous wear of placebo socks for 2 weeks (separated by a 2-week washout period)
* Arm B: Continuous wear of placebo socks for 2 weeks, followed by continuous wear of Voxx Human Performance Technology Socks for 2 weeks (separated by a 2-week washout period)

Patients will be evaluated at three time points using an objective neuropathy assessment as well as self-report questionnaires assessing chemotherapy-induced peripheral neuropathy, quality of life, and cancer-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer, stage 1-4.
* Completed taxane- or platinum-based chemotherapy, vinca alkaloids, or bortezomib at least three months (90 days) ago. Current use of anti-estrogen therapy, Herceptin, or PARP inhibitors is okay.
* Clinical diagnosis of chemotherapy-induced peripheral neuropathy by clinician. This will be based on symptom history (paresthesias, dysesthesias, allodynia), loss of deep tendon reflexes, decreased vibratory sensation, or the presence of symmetrical stocking-glove numbness or paresthesias beginning after neurotoxic chemotherapy.
* Self-reported average neuropathic pain score of at least 4 on a 10-point scale over the past 1 month.
* Age ≥ 18 years
* Concomitant use of analgesics is permitted if the dose has been stable for at least 2 weeks prior to study enrollment (no new analgesics have been added, discontinued, or changed in the 2 weeks prior to randomization).
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Syphilis, alcoholic neuropathy, diabetic neuropathy, neurological disorders, brain injury, or stroke, as assessed by the treating physician.
* Neuropathy related to abnormal thyroid stimulating hormone or cobalamin levels as assessed by treating physician.
* Current severe depression, suicidal ideation, bipolar disease, alcohol abuse, or major eating disorder, as assessed by the treating physician.
* Currently participating in another chemotherapy-induced peripheral neuropathy-targeted program or trial.
* Participated in a non-pharmacologic therapy specifically for the treatment of chemotherapy-induced peripheral neuropathy, including Scrambler Therapy, mindfulness meditation, or other mind-body activities within 14 days (2 weeks) prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cedars Sinai Medical Center, Los Angeles, California
  - CS Cancer at the Hunt Cancer Center, Torrance, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Voxx Socks Followed by Placebo Socks: Continuous wear of Voxx Human Performance Technology Socks for 2 weeks, followed by continuous wear of placebo socks for 2 weeks (separated by a 2-week washout period) Voxx Human Performance Technology Socks: Voxx Human Performance Technology Socks are commercially-available socks that are drug and electrical free. The Voxx Human Performance Technology proprietary pattern is woven into a sock that is made of 70% cotton, 25% polyester, 3% spandex, and 2% nylon.
  Prior to the 2-week treatment window, patients will be provided with 6 pairs of Voxx Human Performance Technology socks. Patients will be asked to wear the socks continuously during both waking and sleeping hours, except when showering, bathing, or swimming.
  Placebo Socks: Placebo socks are identical to the Voxx Human Performance Technology socks but do not include the Voxx Human Performance Technology pattern woven into the sock. Placebo socks are made of the same fabric as Voxx Human Performance Technology socks and are drug and electrical free.
  Prior to the 2-week treatment window, patients will be provided with 6 pairs of placebo socks. Patients will be asked to wear the socks continuously during both waking and sleeping hours, except when showering, bathing, or swimming.
- Arm B: Placebo Socks Followed by Voxx Socks: Continuous wear of placebo socks for 2 weeks, followed by continuous wear of Voxx Human Performance Technology Socks for 2 weeks (separated by a 2-week washout period) Voxx Human Performance Technology Socks: Voxx Human Performance Technology Socks are commercially-available socks that are drug and electrical free. The Voxx Human Performance Technology proprietary pattern is woven into a sock that is made of 70% cotton, 25% polyester, 3% spandex, and 2% nylon.
  Prior to the 2-week treatment window, patients will be provided with 6 pairs of Voxx Human Performance Technology socks. Patients will be asked to wear the socks continuously during both waking and sleeping hours, except when showering, bathing, or swimming.
  Placebo Socks: Placebo socks are identical to the Voxx Human Performance Technology socks but do not include the Voxx Human Performance Technology pattern woven into the sock. Placebo socks are made of the same fabric as Voxx Human Performance Technology socks and are drug and electrical free.
  Prior to the 2-week treatment window, patients will be provided with 6 pairs of placebo socks. Patients will be asked to wear the socks continuously during both waking and sleeping hours, except when showering, bathing, or swimming.
Period: First 2 Week
Arm/Group | Arm A: Voxx Socks Followed by Placebo Socks | Arm B: Placebo Socks Followed by Voxx Socks
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Second 2 Week
Arm/Group | Arm A: Voxx Socks Followed by Placebo Socks | Arm B: Placebo Socks Followed by Voxx Socks
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Voxx Socks Followed by Placebo Socks | Arm B: Placebo Socks Followed by Voxx Socks | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.28571 (16.44304) | 59.85714 (10.91123) | 59.071429 (13.716518)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 14 | 10 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 6 | 8 | 14
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Subjective Measurement of Chemotherapy-induced Peripheral Neuropathy
Description: Impact on chemotherapy-induced peripheral neuropathy will be subjectively measured by changes in scores on the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity Subscale. The minimum value is 0 and maximum value is 44, and a lower score means a better outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Voxx Human Performance Technology Socks: Continuous wear of Voxx Human Performance Technology Socks for 2 weeks
  Voxx Human Performance Technology Socks: Voxx Human Performance Technology Socks are commercially-available socks that are drug and electrical free. The Voxx Human Performance Technology proprietary pattern is woven into a sock that is made of 70% cotton, 25% polyester, 3% spandex, and 2% nylon.
  Prior to the 2-week treatment window, patients will be provided with 6 pairs of Voxx Human Performance Technology socks. Patients will be asked to wear the socks continuously during both waking and sleeping hours, except when showering, bathing, or swimming.
- Placebo Socks: Continuous wear of placebo socks for 2 weeks
  Placebo Socks: Placebo socks are identical to the Voxx Human Performance Technology socks but do not include the Voxx Human Performance Technology pattern woven into the sock. Placebo socks are made of the same fabric as Voxx Human Performance Technology socks and are drug and electrical free.
  Prior to the 2-week treatment window, patients will be provided with 6 pairs of placebo socks. Patients will be asked to wear the socks continuously during both waking and sleeping hours, except when showering, bathing, or swimming.
Arm/Group | Voxx Human Performance Technology Socks | Placebo Socks
Number analyzed (Participants) | 28 | 28
score on a scale | 27.32 (8.03) | 27.94 (8.72)

2. Secondary Outcome: Change in Objective Measurement of Chemotherapy-induced Peripheral Neuropathy (Score on the Modified Total Neuropathy Scale)
Description: Impact on chemotherapy-induced peripheral neuropathy will be objectively measured by changes in scores on the Total Neuropathy Scale clinical. The minimum value is 0 and maximum value is 28, and a lower score means a better outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo Socks: Continuous wear of placebo socks for 2 weeks,
  Placebo Socks: Placebo socks are identical to the Voxx Human Performance Technology socks but do not include the Voxx Human Performance Technology pattern woven into the sock. Placebo socks are made of the same fabric as Voxx Human Performance Technology socks and are drug and electrical free.
  Prior to the 2-week treatment window, patients will be provided with 6 pairs of placebo socks. Patients will be asked to wear the socks continuously during both waking and sleeping hours, except when showering, bathing, or swimming.
Arm/Group | Voxx Human Performance Technology Socks | Placebo Socks
Number analyzed (Participants) | 27 | 26
score on a scale | 8.22 (2.36) | 8.88 (3.13)

3. Secondary Outcome: Change in Objective Measurement of Chemotherapy-induced Peripheral Neuropathy (Score on the Timed Up and Go Test)
Description: Impact on chemotherapy-induced peripheral neuropathy will be objectively measured by changes in scores on the Timed Up and Go test.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Voxx Human Performance Technology Socks | Placebo Socks
Number analyzed (Participants) | 27 | 27
seconds | 10.19 (2.96) | 10.55 (3.02)

4. Secondary Outcome: Change in Quality of Life Measurement
Description: Impact on quality of life will be measured by the changes in scores on the Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29). PROMIS-29 is a collection of short form instruments which encompass PROMIS domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social and activities) in addition to a single item assessing pain intensity. The PROMIS 29 contains 4 items per domain plus one pain intensity item, totaling 29 items. Each domain is scored separately. For all domains (besides pain intensity) the raw score lies between 4 to 20. The PROMIS-29 uses a T-score metric to score its domains, with a mean of 50 and a standard deviation of 10, where higher scores indicate better health or less of the concept being measured.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voxx Human Performance Technology Socks | Placebo Socks
Number analyzed (Participants) | 28 | 28
score on a scale
  Physical Function | 43.19 (8.29) | 42.66 (8.94)
  Anxiety | 52.86 (9.36) | 52.76 (9.13)
  Depression | 50.04 (9.29) | 49.63 (8.93)
  Fatigue | 52.18 (9.65) | 53.94 (11.12)
  Sleep Disturbance | 57.03 (2.57) | 56.76 (2.67)
  Pain Interference | 57.75 (8.97) | 58.2 (8.69)
  Ability to participate in social and activities | 49.86 (8.78) | 49.11 (10.41)

5. Secondary Outcome: Change in Cancer-related Symptom Experience
Description: Impact on cancer-related symptom experience will be measured by changes in scores on the Edmonton Symptom Assessment Scale. The minimum value is 0 and maximum value is 100, and a lower score means a better outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voxx Human Performance Technology Socks | Placebo Socks
Number analyzed (Participants) | 28 | 28
score on a scale | 26.39 (17.89) | 27.61 (18.1)

6. Secondary Outcome: Feasibility of Voxx Socks Use
Description: Feasibility will be measured by the number of hours the socks are worn, as recorded in the patient's daily sock diary.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Voxx Human Performance Technology Socks | Placebo Socks
Number analyzed (Participants) | 25 | 25
hours/day | 17.31615 (6.463149) | 16.65153 (6.011369)

ADVERSE EVENTS:
Time Frame: from the start of treatment until 30 days following the end of treatment or until initiation of a new anticancer therapy (whichever occurs first)
Groups:
- Placebo Socks: Continuous wear of placebo socks for 2 weeks
  Voxx Human Performance Technology Socks: Voxx Human Performance Technology Socks are commercially-available socks that are drug and electrical free. The Voxx Human Performance Technology proprietary pattern is woven into a sock that is made of 70% cotton, 25% polyester, 3% spandex, and 2% nylon.
  Prior to the 2-week treatment window, patients will be provided with 6 pairs of Voxx Human Performance Technology socks. Patients will be asked to wear the socks continuously during both waking and sleeping hours, except when showering, bathing, or swimming.
Arm/Group | Voxx Human Performance Technology Socks | Placebo Socks
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 3/28 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voxx Human Performance Technology Socks (N=28) | Placebo Socks (N=28)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1)
Other - Skin Iritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT04403802/Prot_SAP_002.pdf
  • Informed Consent Form (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/02/NCT04403802/ICF_001.pdf